CLINICAL TRIAL: NCT03071432
Title: QUANtification of Cardiovascular Autonomic Neuropathy (CAN) and the Effects of Anaesthesia on Haemodynamics and Cerebral Perfusion
Acronym: QUANCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Principal Investigator, B Preckel, Professor in anesthesiology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC2016_116
Record Dates: First submitted 2017-02-20; First posted 2017-03-07 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Non-diabetic patients, n=15 Diabetic patients with cardiovascular autonomic neuropathy, n=15 Diabetic patients without cardiovascular autonomic neuropathy, n=15
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-diabetic patients (Active Comparator): Study interventions include a medical history and short physical examination as well as autonomic function tests and cerebral autoregulation tests on the day before surgery. In addition we determine CO2 sensitivity of the cerebral vasculature by three minutes hyperventilation and three minutes CO2 rebreathing. Perioperatively, continuous measurement of heart rate, blood pressure, stroke volume and cardiac output is aquired using the ccNexfin monitor, a non-invasive device using a single finger cuff. Continuous monitoring of cerebral perfusion parameters using transcranial Doppler ultrasound (TCD) of the middle cerebral artery (MCA) and cerebral oxygenation using near-infrared-spectroscopy (NIRS) will be obtained. BRS and condition of CA will be determined preoperatively during autonomic function testing (see below) and 30 minutes after induction of anaesthesia.
  Interventions: Diagnostic Test: Paced breathing at 6, 10 and 15 breaths per minute
- Diabetic patients with cardiovascular autonomic neuropathy (Active Comparator): Study interventions include a medical history and short physical examination as well as autonomic function tests and cerebral autoregulation tests on the day before surgery. In addition we determine CO2 sensitivity of the cerebral vasculature by three minutes hyperventilation and three minutes CO2 rebreathing. Perioperatively, continuous measurement of heart rate, blood pressure, stroke volume and cardiac output is aquired using the ccNexfin monitor, a non-invasive device using a single finger cuff. Continuous monitoring of cerebral perfusion parameters using transcranial Doppler ultrasound (TCD) of the middle cerebral artery (MCA) and cerebral oxygenation using near-infrared-spectroscopy (NIRS) will be obtained. BRS and condition of CA will be determined preoperatively during autonomic function testing (see below) and 30 minutes after induction of anaesthesia.
  Interventions: Diagnostic Test: Paced breathing at 6, 10 and 15 breaths per minute
- Diabetic patients without cardiovascular autonomic neuropathy (Active Comparator): Study interventions include a medical history and short physical examination as well as autonomic function tests and cerebral autoregulation tests on the day before surgery. In addition we determine CO2 sensitivity of the cerebral vasculature by three minutes hyperventilation and three minutes CO2 rebreathing. Perioperatively, continuous measurement of heart rate, blood pressure, stroke volume and cardiac output is aquired using the ccNexfin monitor, a non-invasive device using a single finger cuff. Continuous monitoring of cerebral perfusion parameters using transcranial Doppler ultrasound (TCD) of the middle cerebral artery (MCA) and cerebral oxygenation using near-infrared-spectroscopy (NIRS) will be obtained. BRS and condition of CA will be determined preoperatively during autonomic function testing (see below) and 30 minutes after induction of anaesthesia.
  Interventions: Diagnostic Test: Paced breathing at 6, 10 and 15 breaths per minute

INTERVENTIONS:
Diagnostic Test: Paced breathing at 6, 10 and 15 breaths per minute

SUMMARY:
Rationale: Complications of chronic hyperglycaemia associated with Diabetes Mellitus type 2 (DM2) include macro- and microvascular angiopathy. Cerebral Autoregulation (CA), the capability of the brain to maintain constant cerebral blood flow (CBF) despite changes in blood pressure, is impaired early in DM2 implicating that CBF becomes dependent on blood pressure. In addition, 20-60% of all patients with DM2 suffers from cardiovascular autonomic neuropathy (CAN) resulting in more unstable blood pressure regulation. In patients without DM2 or CAN, induction of anaesthesia results in slightly decreased blood pressure, but cerebral perfusion is maintained through CA. In contrast, patients with DM2 and CAN may display greater reductions in blood pressure and cerebral perfusion may become jeopardized due to impaired CA. This could be an explanation for the increased incidence of stroke in patients with DM2.

Objective:

1. To study whether peri-operative haemodynamics fluctuate more in patients with DM2 and CAN.
2. To study whether CAN further worsens cerebral perfusion in addition to impaired CA.

Study design: Prospective, observational cohort trial. Study population: A total of 45 patients, 30 with DM2 and 15 healthy controls scheduled for elective, non-cardiothoracic surgery under general anesthesia and age 18 years and above will be included in the study. After inclusion, DM2-patients will be categorized in two groups (both 15 patients): patients with and patients without CAN. Given the prevalence of 20-60% CAN, we plan to screen at most 100 patients and include 15 patients in each study group.

Intervention (if applicable):

1. PRE-operative: chart review, short physical examination, autonomic function tests to determine the presence of CAN. These tests are simple physiological tests that can be performed on a regular ward and involve a Vasalva manoeuvre, 3 minute paced breathing with a frequency of 6·min-1 and tests for orthostatic hypotension. Also, we test the sensitivity of the cerebral vasculature to CO2 by measuring during one-minute hyperventilation and one minute CO2-rebreathing. Continuous blood pressure monitoring will be obtained using ccNexfin, a non-invasive monitor that comprises a single inflatable finger cuff. Cerebral perfusion will be assessed non-invasively using transcranial Doppler attached with a headband to the temporal skin area and (non-invasive) measurement of cerebral oxygenation using near-infrared spectroscopy (NIRS).
2. INTRA-operative: we repeat the 3 minute paced breathing test and the CO2-reactivity test.

Main study parameters/endpoints: Between group difference in haemodynamic parameters and cerebral perfusion parameters.

ELIGIBILITY:
Inclusion criteria:

* Willing and able to give written informed consent
* Scheduled for elective, non-cardiothoracic surgery under general anesthesia
* Age 18 years and above

Exclusion criteria:

* Day case surgery
* laparoscopic procedure
* DM type 1
* Parkinson's disease
* uncontrolled cardiac arrhythmia
* Pure autonomic failure (formerly called idiopathic orthostatic hypotension)
* Multiple system atrophy with autonomic failure (formerly called Shy-Drager syndrome)
* Addison's disease and hypopituitarism
* pheochromocytoma
* peripheral autonomic neuropathy (e.g., amyloid neuropathy, idiopathic autonomic neuropathy)
* known cardiomyopathy
* extreme left ventricle hypertrophy or ejection fraction < 30%
* proven or suspected allergy for any of the medication used during induction of anaesthesia
* malignant hyperthermia
* unability to record transcranial doppler ultrasound due to anatomical variance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in baroreflex sensitivty after induction of anesthesia | Pre-operative versus Intra-operative
  Baroreflex sensitivity (BRS; expressed as ms change in R-R-interval per mmHg blood pressure change) can be seen as a measure of hemodynamic homeostatic control. We calculate BRS preoperatively (baseline) and compare it to intra-operative values (after induction of anesthesia).
Change from baseline in dynamic cerebral autoregulation after induction of anesthesia | Pre-operative versus Intra-operative
  Dynamic Cerabral Autoregulation (dCA; expressed as MCAVmean-to-MAP phase lead) can be seen as the ability of the brain to compensate for blood pressure changes. We calculate dCA pre-operatively (baseline) and compare it to intra-operative values (after induction of anesthesia).

SECONDARY OUTCOMES:
Clinical outcome | Intra-operative till 30 days postoperative
  The relationship between autonomic function tests and clinical outcome during 30-postoperative days (observational). Outcome measures include frequency of all adverse and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sperna Weiland NH, Hermanides J, van der Ster BJP, Hollmann MW, Preckel B, Stok WJ, van Lieshout JJ, Immink RV. Sevoflurane based anaesthesia does not affect already impaired cerebral autoregulation in patients with type 2 diabetes mellitus. Br J Anaesth. 2018 Dec;121(6):1298-1307. doi: 10.1016/j.bja.2018.07.037. Epub 2018 Sep 6. PMID 30442257
- [Derived] Sperna Weiland NH, Hermanides J, Hollmann MW, Preckel B, Stok WJ, van Lieshout JJ, Immink RV. Novel method for intraoperative assessment of cerebral autoregulation by paced breathing. Br J Anaesth. 2017 Dec 1;119(6):1141-1149. doi: 10.1093/bja/aex333. PMID 29028933